CLINICAL TRIAL: NCT04007341
Title: Effect of Dexmedetomidine on the Inflammatory Response in Patients Undergoing Lung Resection Surgery
Brief Title: Effect of Dexmedetomidine on the Inflammatory Response After One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Wonjung Hwang, Assistant professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC16MISI0042
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline group (No Intervention): Patients in the saline group were infused with an identical volume of normal saline.
- Dexmedetomidine group (Experimental): Patients in the dexmedetomidine group were infused with a loading dose of dexmedetomidine (1.0 mcg/kg over 10 min) and were thereafter infused at a rate of 0.5 mg/kg/h.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The study drug for each group was administered from the time immediately after induction of anesthesia until the end of the surgery.
  Arms: Dexmedetomidine group

SUMMARY:
The postoperative inflammatory response is significant in lung resection surgery because of major operation and one-lung ventilation. Dexmedetomidine has been shown to reduce pro-inflammatory cytokine levels and improve clinical outcomes. The aim of this study was to determine the effects of dexmedetomidine on inflammatory responses after lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective video-assisted thoracoscopic surgery (VATS) lobectomy
* 20 < age < 75
* American Society of Anesthesiologists (ASA) classification I~II

Exclusion Criteria:

* preoperative inflammation (CRP>10ng/#, WBC>10,000/mm3, body temperature >38#)
* steroid administration within 1 month
* hematologic / autoimmune disease
* congestive heart failure (NYHA class III~IV) or significant arrhythmia
* severe obstructive / restrictive pulmonary disease
* previous history of thoracic surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-29 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Interleukin (IL)-6 | 24 hours after surgery
  Blood samples were collected from the antecubital vein

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea